CLINICAL TRIAL: NCT06297460
Title: Adaptation of the Systems Training for Emotional Predictability & Problem Solving (STEPPS) Program for Addressing Emotional Dysregulation and Self-harming Behaviors in Penitentiary Centers in Catalonia
Brief Title: Adaptation of STEPPS Program for Addressing Emotional Dysregulation and Self-harming Behaviors in Penitentiary Centers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Centre d'Estudis i Formació Especialtzada Generalitat de Catalunya (Unknown)
Responsible Party: Principal Investigator, Rosa Lorente, Senior Research Technical Staff, Universitat Jaume I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEPPSPENITENTIARY
Record Dates: First submitted 2024-01-08; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Self Harm
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEPPS program (Experimental): The only condition is the experimental one. Participants receive the STEPPS program
  Interventions: Behavioral: Systems Training for Emotional Predictability & Problem Solving (STEPPS)

INTERVENTIONS:
Behavioral: Systems Training for Emotional Predictability & Problem Solving (STEPPS) — STEPPS is based on a cognitive-behavioral and skills training approach divided into three major components. The first component (sessions: 1-2) teaches participants to replace misconceptions about the presented issues with greater awareness of thoughts, feelings, and behaviors that characterize them. It also helps them identify their own thought patterns driving their behaviors. The second (sessions 3-12) teaches skills to more effectively manage the cognitive and emotional effects of the issues, such as distancing, communication, challenging, distraction, and problem-solving. The third component (sessions 13-19) teaches behavioral skills where participants are encouraged to master habits of healthy eating, sleep hygiene, regular exercise, leisure activities, health monitoring, self-harm prevention, and interpersonal effectiveness. The therapeutic objectives of the three blocks are awareness of illness (1), emotional regulation (2), and behavioral regulation (3).

SUMMARY:
The overall objective of this study is to assess the feasibility, within the Penitentiary Centers of Catalonia, of adapting the STEPPS program for addressing and preventing emotional dysregulation and self-harming behaviors through an implementation study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women deprived of liberty serving sentences in a penitentiary center in Catalonia.
* Presence of self-harming behaviors.
* Sufficient understanding and proficiency in Spanish to participate in the STEPPS program.
* Sufficient cognitive competence for study participation.
* Mental capacity to provide informed consent.

Exclusion Criteria:

* Inmates under security measures or classified in the first degree of treatment.
* Inmates with language difficulties.
* Presence of severe pathologies that may hinder study participation.
* Inmates with the possibility of imminent release, impending transfers to other penitentiary centers, or pending trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Level of emotional and behavioral disregulation of patients | Pre-intervention and inmediately after the intervention
  Using the Longitudinal assessment of the severity of emotional and behavioral dysregulation (Borderline Evaluation of Severity Over Time, BEST) (Blum et al., 2002), a 15-item questionnaire with a 5-point Likert scale (1= none/very mild; 5= extremely) that assesses three areas: the intensity of thoughts and emotions, and negative and positive behaviors.

SECONDARY OUTCOMES:
Type and levels of impulsivity of patients | Pre-intervention and inmediately after the intervention
  The Barratt Impulsiveness Scale (BIS) (Barratt, 1959) is a self-report questionnaire designed to assess impulsiveness in different areas. It consists of 30 items that are scored on a 4-point scale (from rarely or never (1) to always or almost always (4)). The scale measures three aspects of impulsiveness: Attentional Impulsiveness, Motor Impulsiveness, and Non-Planning Impulsiveness.
Suicide risk of patients | Pre-intervention and inmediately after the intervention
  Using the Beck Suicidal Intent Scale (SIS) (Beck et al., 1979) it is assessed the characteristics and likelihood of a suicide attempt in the present and the past. It addresses circumstances during the attempt, attitudes towards life and death, thoughts before, during, and after the attempt, and substance use. The questionnaire consists of 20 items rated on a 3-point scale (0 to 2).
Self-injury frequency, typology and funcionality of patients | Pre-intervention and inmediately after the intervention
  Through Inventory of Statements About Self-injury (ISAS) (Klonsky & Glenn, 2009), a questionnaire that explores self-injurious behaviors and is divided into two sections. The first section evaluates the presence and frequency of 13 different types of self-injuries, and the second section assesses the functionality of self-injurious behaviors on a 3-point Likert scale.
Degree of hopeless of patients | Pre-intervention and inmediately after the intervention
  Using Beck Hopeless Scale (BHS) (Beck et al., 1974), a 20-item true/false scale that assesses individuals' feelings of hopelessness. In this case, it evaluates three aspects of hopelessness: 1. A person's expectations about life; 2. Their feelings about the future, and 3. The loss of motivation.
Perceived level of feasibility by professionals | Pre-intervention and inmediately after the intervention
  Feasibility is measured with the Feasibility of Intervention Measure (FIM) (Weiner et al., 2017), a measure that encompasses four items designed to measure the feasibility of the intervention, indicating the extent to which the intervention can be successfully executed within the system, using a 5-point Likert scale.
Perceived level of acceptability of the intervention by professionals | Pre-intervention and inmediately after the intervention
  The Acceptability of Intervention Measure (AIM) (Weiner et al., 2017) assesses acceptability based on stakeholders' perceptions of the intervention's utility or satisfaction across four items on a 5-point Likert scale.
Satisfaction of the intervention by patients | Pre-intervention and inmediately after the intervention
  The Client Satisfaction Questionnaire (CSQ) (Attkisson & Zwick, 1982; Larsen et al., 1979) is an eight-item questionnaire that assesses participants' overall satisfaction with the intervention received on a 4-point scale.
Perceived level of adequacy by professionals | Pre-intervention and inmediately after the intervention
  Intervention Appropriateness Measurement (IAM) (Weiner et al., 2017) comprises four 5-point Likert scale items designed to explore the adequacy of the intervention, considering its perceived relevance or compatibility in the given context.
Barriers and facilitators detected by professionals that are influencing the implementation process - Quantitative information | Pre-intervention and inmediately after the intervention
  Quantitative data about barriers and facilitators is gathered thrhough closed-open questionnaire was developed following CFIR guidelines (Damschroder et al., 2009), with reference to the study conducted by Hadjistavropoulos and colleagues (2017). The final questionnaire comprised 41 items rated on a 5-point Likert scale (ranging from 1, strongly disagree, to 5, strongly agree), assessing: Intervention Characteristics (7 items), Outer Context (5 items), Inner Setting (14 items), Characteristics of Individuals (8 items), and Implementation Process (7 items).
Level of burnout of professionals | Pre-intervention and inmediately after the intervention
  Using the Copenhagen Burnout Inventory (CBI) (Kristensen et al., 2005), a 19-item questionnaire on a 5-point Likert scale that measures burnout syndrome, differentiating three sub-dimensions: personal burnout, work-related burnout, and user-related burnout.

OTHER OUTCOMES:
Barriers and facilitators detected by professionals that are influencing the implementation process - Qualitative information | Inmediately after the intervention
  Semi-structured interviews conducted to professionals guided by Consolidated Framework for Implementation Research (CFIR) (Damschroder et al., 2009).
  To guide the development of these analyses, the CFIR served as a framework, assisting in semi-structured interviews and formulating relevant questions based on the five domains that influence the implementation process: (1) Intervention Characteristics, (2) Outer Setting, (3) Inner Setting, (4) Characteristics of Individuals, and (5) Implementation Process (25,33).

CONTACTS AND LOCATIONS:
Locations (1):
- Rosa, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black DW, Blum N, Eichinger L, McCormick B, Allen J, Sieleni B. STEPPS: Systems Training for Emotional Predictability and Problem Solving in women offenders with borderline personality disorder in prison--a pilot study. CNS Spectr. 2008 Oct;13(10):881-6. doi: 10.1017/s1092852900016989. PMID 18955943
- [Background] Black DW, Blum N, McCormick B, Allen J. Systems Training for Emotional Predictability and Problem Solving (STEPPS) group treatment for offenders with borderline personality disorder. J Nerv Ment Dis. 2013 Feb;201(2):124-9. doi: 10.1097/NMD.0b013e31827f6435. PMID 23364121
- [Background] Arnau F, Garcia-Guerrero J, Benito A, Vera-Remartinez EJ, Baquero A, Haro G. Sociodemographic, Clinical, and Therapeutic Aspects of Penitentiary Psychiatric Consultation: Toward Integration Into the General Mental Health Services. J Forensic Sci. 2020 Jan;65(1):160-165. doi: 10.1111/1556-4029.14137. Epub 2019 Jul 25. PMID 31343744
- [Background] Brennan CA, Crosby H, Sass C, Farley KL, Bryant LD, Rodriquez-Lopez R, Romeu D, Mitchell E, House AO, Guthrie E. What helps people to reduce or stop self-harm? A systematic review and meta-synthesis of first-hand accounts. J Public Health (Oxf). 2023 Mar 14;45(1):154-161. doi: 10.1093/pubmed/fdac022. PMID 35211734
- [Derived] Lorente-Catala R, Jaen I, Busca-Huertas X, Framis B, Garcia-Palacios A. Implementation of the STEPPS program for the treatment of self-harm behaviors in Catalonia's prisons: barriers and facilitators. BMC Public Health. 2025 Jan 30;25(1):378. doi: 10.1186/s12889-025-21519-8. PMID 39885488
- [Derived] Lorente-Catala R, Jaen I, Busca-Huertas X, Framis B, Garcia-Palacios A. Treating self-harm behaviors in prisons: implementation of the STEPPS program. BMC Psychol. 2025 Jan 16;13(1):43. doi: 10.1186/s40359-024-02342-z. PMID 39819704